CLINICAL TRIAL: NCT06607549
Title: A Phase 1 Study of Loncastuximab Tesirine and Rituximab Following Stereotactic Radiosurgery (SRS) in Patients With Primary and Secondary Central Nervous System Lymphomas
Brief Title: Loncastuximab Tesirine and Rituximab Following Stereotactic Radiosurgery in Patients With Central Nervous System Lymphomas (SOLAR)
Acronym: SOLAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI181535
Record Dates: First submitted 2024-09-13; First posted 2024-09-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Central Nervous System Lymphoma
MeSH Terms: interventions — loncastuximab tesirine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: All Patients (Experimental): This study has two main goals:
  Goal 1: The study will investigate the safety and tolerability of loncastuximab tesirine and rituximab (lonca-R).
  Goal 2: The study will determine the maximum tolerated dose of lonca-R.
  Interventions: Drug: Loncastuximab tesirine and rituximab (Lonca-R)

INTERVENTIONS:
Drug: Loncastuximab tesirine and rituximab (Lonca-R) — Patients will receive stereotactic radiosurgery (SRS) followed by a brain MRI approx. 3 weeks after SRS. This will be followed by loncastuximab tesirine and rituximab administered intravenously for a total of 6 cycles (every 21 days).

SUMMARY:
The purpose of this clinical trial is to learn if drugs loncastuximab tesirine and rituximab (lonca-R) after stereotactic radiosurgery are safe and effective for treatment of central nervous system lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years
* ECOG Performance Status ≤ 3
* Histologically confirmed primary CNS lymphoma or secondary diffuse large B-cell lymphoma (DLBCL) with CNS involvement with either:

  * Relapsed or refractory disease with at least 1 prior therapy OR
  * Ineligible for high-dose methotrexate-based therapy as determined by the treating physician, including previously untreated patients. Examples of medical conditions for which a patient could be considered ineligible for high-dose methotrexate include but not limited to renal impairment, liver disease, heart failure.

    * Note: For patients with a history of histologically documented systemic DLBCL with CNS relapse, a biopsy of the CNS lesion is recommended but not required.
* Must be a candidate for SRS. Lesion size must be < 6 cm and the number of lesions must be < 10.
* Must have evaluable disease. This includes radiographic evidence of parenchymal disease or parenchymal disease and disease detected in the CSF.

  * Patients with vitreous or retinal involvement alone are not eligible.
  * Patients with leptomeningeal disease or spinal cord disease are not eligible.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count ≥ 1000 cells/mm3 (1.00 x 109/L) independent of G-CSF support (i.e. no G-CSF within the past 3 days) unless there is documented bone marrow involvement.
    * Platelet count ≥ 75,000 cells/mm3 (75 x 109/L) independent of transfusion support (i.e. no transfusion within the past 3 days) unless there is documented bone marrow involvement.
    * Hemoglobin ≥ 8 g/dL (≥ 80 g/L) independent of transfusion support (i.e. no transfusion within the past 3 days) unless there is documented bone marrow involvement.
  * Hepatic:

    ---Total bilirubin ≤ 2.0 mg/dL (unless bilirubin rise is due to Gilbert's syndrome), if total bilirubin is > 2.0 mg/dL, the subject is eligible for the study if the direct bilirubin is normal; transaminases (AST/ALT) ≤2.5 x upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:

      * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
      * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
* For subjects of childbearing potential: Negative pregnancy test or evidence of permanent surgical sterilization. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago
* Female participants of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.1 until 10 months after last dose of loncastuximab tesirine and 12 months after the last dose of rituximab. Male participants with female partners of childbearing potential must agree to use a highly effective method of contraception when sexually active until 7 months after the last dose of loncastuximab tesirine.
* Provide written informed consent and comply with the study protocol as judged by the Investigator. Of note, if the subject has an impairment that prevents him/her from providing consent, the site may follow approved institutional procedures for obtaining consent. The investigator should document when a potential or current participant lacks decision-making capacity and thus requires an LAR to provide consent.

Exclusion Criteria:

* Concurrent use of other approved or investigational antineoplastic agents (with the exception of corticosteroids).
* History of intracranial hemorrhage or clinically significant stroke within 6 months prior to enrollment
* History of prior radiation to the CNS.
* Significant medical diseases or conditions, as assessed by the investigator, that would substantially increase the risk-to-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction in the past 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, severely immunocompromised state, and congestive heart failure, New York Heart Association Class III-IV.
* Known bleeding diathesis (e.g., von Willebrand's disease), hemophilia, or active bleeding.
* Known Human immunodeficiency virus (HIV) infection.
* Prior allogeneic stem cell transplant (autologous stem cell transplant is NOT an exclusion).
* Prior exposure to loncastuximab tesirine
* Chemotherapy or targeted small molecule therapy (or other therapy for CNS lymphoma) within 3 weeks prior to the first day of study treatment (or 5 half-lives (whichever is shorter), or 2 weeks prior to the first day of study treatment for monoclonal antibodies.
* The patient must have recovered to baseline or ≤ grade 1 from prior toxicities of therapy with the exception of alopecia and myelosuppression provided lab criteria met. Recovery to ≤ grade 2 neuropathy is permitted.
* Cellular therapy within 8 weeks.
* Presence of clinically significant pericardial or pleural effusions, or third space fluid accumulations (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
* Congenital long QT syndrome or a corrected QT measure (QTc) interval of >480 ms at screening (unless secondary to pacemaker or bundle branch block).
* Known history of hypersensitivity to CD19 antibody and/or, components of study medication.
* All subjects must be screened for hepatitis B and C. Patients with evidence of active hepatitis B infection, based on positive surface antigen or Hepatitis B DNA PCR are excluded. Patients who are Hepatitis B core antibody positive must take prophylaxis with entecavir or equivalent and be willing to undergo monthly Hepatitis B DNA PCR testing. Subjects with active Hep C patients may be enrolled if other parameters precluding hepatic impairment are met and they are not undergoing active therapy for hepatitis C.
* Active systemic bacterial, viral, fungal, or other infection requiring systemic treatment at time of screening.
* Subjects with chronic liver disease with hepatic impairment Child-Pugh class C
* Pregnant or lactating or intending to become pregnant during the study.
* Patients diagnosed with another malignancy within three years or with any evidence of residual prior malignant disease (except nonmelanoma skin cancer, non-metastatic prostate cancer, in situ cervical cancer, or ductal or lobular carcinoma in situ). Patients meeting this exclusion criteria may be enrolled after approval from study PI.
* Unable to tolerate corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
A safe and tolerable dose of lonca-R following SRS in patients with CNS lymphoma who have relapsed disease or are untreated and not candidates for HDMTX-based therapy. | 5 years
  Maximum Tolerated Dose (MTD): MTD is defined as the highest dose under consideration that has an estimated DLT probability below 25% based upon the Bayesian optimal interval design. The MTD will be decided based on the BOIN decision rules set for phase 1a portion of the study.

SECONDARY OUTCOMES:
To assess best overall response rate (ORR) following lonca-R | 6 months
  To evaluate the preliminary efficacy (ORR) of lonca-R following SRS in patients with CNS lymphoma who have relapsed disease or are untreated and not candidates for HDMTX-based therapy.
To assess best complete response (CR) rate following lonca-R. | 6 months
  To evaluate the preliminary efficacy (complete response rate) of lonca-R following SRS in patients with CNS lymphoma who have relapsed disease or are untreated and not candidates for HDMTX-based therapy.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment. | 5 years
  To determine the safety and tolerability of lonca-R following SRS in patients with CNS lymphoma who have relapsed disease or are untreated and not candidates for HDMTX-based therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Narendranath Epperla, MD, MS, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No